CLINICAL TRIAL: NCT03108170
Title: Digital Perineal Massage and Pelvic Floor Muscle Exercise as an Antenatal Program for Prevention of Perineal Trauma in Elderly Women, a Randomized Controlled Trial
Brief Title: Digital Perineal Massage and Pelvic Floor Muscle Exercise During Pregnancy for Prevention of Perineal Laceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3644
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Delivery; Injury, Maternal
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 programs group (Active Comparator): The participants will receive 3 programs.The educational pelvic floor dysfunction prevention program, pelvic floor muscle exercise program and perineal massage program will be educated by an investigator during the participant visit 4 weeks before her duo date
  Interventions: Other: perineal massage program; Other: Pelvic floor muscle exercise program; Other: Educational pelvic floor dysfunction prevention program
- one program group (Active Comparator): The participants will receive one program. That is the educational pelvic floor dysfunction prevention program.The instructions of the program will be given by an investigator once during the participant visit 4 weeks before her duo date.
  Interventions: Other: Educational pelvic floor dysfunction prevention program

INTERVENTIONS:
Other: perineal massage program — The participant will perform digital massage of her perineal area 5 minutes daily starting four weeks before delivery till her actual labour day
  Arms: 3 programs group
Other: Pelvic floor muscle exercise program — The participant will perform pelvic floor muscle exercise daily starting four weeks before delivery till her actual labour day
  Arms: 3 programs group
Other: Educational pelvic floor dysfunction prevention program — This educational pelvic floor dysfunction prevention program includes instructions about: control of her weight, adequate cleaning for the perineal area, adequate fluid intake, smoking cessation, right posture and frequency of micturition and adequate ingestion of fiber to avoid constipation

SUMMARY:
Pregnant participants will be recruited at the obstetrics outpatient clinic during their visits 4 weeks before the due date. They are randomized into two groups. The first group will be educated to do digital perineal massage. They will be also educated to do pelvic floor muscle exercises and will receive the usual education program for strengthening the pelvic floor. The second group will receive the usual education program for strengthening the pelvic floor. Occurrence of perineal laceration will be reported at time of delivery.

DETAILED DESCRIPTION:
Pregnant participants will be recruited at the obstetrics outpatient clinic during their visits 4 weeks before the due date. They are randomized into two groups. The first group will be educated to do digital perineal massage. They will be also educated to do pelvic floor muscle exercises and will receive the usual educational pelvic floor dysfunction prevention program for strengthening the pelvic floor. The second group will receive the usual education program for strengthening the pelvic floor. Occurrence of perineal laceration will be reported at time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 35 years old
* Primigravida or multi gravida

Exclusion Criteria:

* History of chronic constipation
* History of chronic cough
* Current or past urinary or anal incontinence
* History of genital prolapse before pregnancy
* History of neuromuscular disorders or connective tissue disorders
* History of medical disorders
* History of preterm or precipitate labour
* History of premature preterm rupture of membranes.
* Genital infections

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who have perineal tears | At 15 minutes from delivery
  Proportion of perineal tears will be assessed by an investigator who will attend the participant delivery

SECONDARY OUTCOMES:
Proportion of participants who need episiotomy at time of delivery | At 15 minutes from delivery
  Proportion of participants who need episiotomy at time of delivery will be assessed by an investigator
Duration of the second stage of labour | At 15 minutes from delivery
  Duration of the second stage of labour will be assessed by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes